CLINICAL TRIAL: NCT01262885
Title: A Randomized, Single Blind, Placebo Controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Oral Doses and Repeat Escalating Oral Doses of GSK2251052 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114470
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Infections, Bacterial
Keywords: pharmacokinetics; tolerability; single dose; antibiotics; repeat dose; GSK2251052; safety
MeSH Terms: conditions — Bacterial Infections | interventions — 3-(aminomethyl)-7-(3-hydroxypropoxy)-1-hydroxy-1,3-dihydro-2,1-benzoxaborole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A Cohort 1 (Experimental): GSK2251052 500 mg (6 subjects), Placebo (1 subject)
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part A Cohort 2 (Experimental): GSK2251052 1000 mg (6 subjects), Placebo (1 subject)
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part A Cohort 3 (Experimental): GSK2251052 2000 mg (6 subjects), Placebo (1 subject)
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part A Cohort 2 - fed (Experimental): GSK2251052 1000 mg (6 subjects), Placebo (1 subject)
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part B Cohort 1 (Experimental): Placebo (3 subjects), GSK2251052 (9 subjects) dose to be determined
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part B Cohort 2 (Experimental): Placebo (3 subjects), GSK2251052 (9 subjects) dose to be determined
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part B Cohort 3 (Experimental): Placebo (3 subjects), GSK2251052 (9 subjects) dose to be determined
  Interventions: Drug: GSK2251052; Drug: Placebo
- Part A Cohort 4 (Experimental): Placebo (1 subject), GSK2251052 (6 subjects) dose to be determined
  Interventions: Drug: GSK2251052; Drug: Placebo

INTERVENTIONS:
Drug: GSK2251052 — 500 mg tablet, dose levels detailed in Arm description
Drug: Placebo — matching placebo tablet

SUMMARY:
GSK2251052 ((S)-3-(aminomethyl)-7-(3-hydroxypropoxy)-1-hydroxy-1,3-dihydro-2,1-benzoxaborole hydrochloride) is a Gram negative antibacterial compound currently in development for the treatment of hospital acquired Gram negative infection (including E. coli, K. pneumoniae, and Enterobacter spp.) This study will be conducted in two (2) parts, with single oral doses being explored in Part A (500, 1000, and 2000 mg) and repeat oral doses (1000 and 2000 mg, b.i.d.) being explored in Part B. Parts A and B will be single-blind, randomized, placebo-controlled, dose-rising studies in healthy subjects to evaluate the safety, tolerability and pharmacokinetics of oral GSK2251052.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin < or = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Abnormal LFT tests may be repeated once at the discretion of the Investigator. If an abnormality is repeated, the subject would not be eligible for inclusion.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with coagulation, reticulocyte, or Hgb values outside the normal range should always be excluded from enrollment.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until at least 90 days post-last dose.
* Body weight > 50 kg and BMI within the range 19 - 32 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTc, QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma, (e.g., for any FTIH where risk of bronchoconstriction is unknown, or compound specific where risk of bronchoconstriction).
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* A history of orthostatic hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2011-08-25 (Actual); Study Completion 2011-08-25 (Actual)

PRIMARY OUTCOMES:
Adverse event reporting, clinical laboratory tests, vital signs, cardiac monitoring, urinalysis, and clinical monitoring/observation. | within 35 days of first dose
Plasma AUC(0-t), AUC(0-inf), Cmax, tmax, t1/2, Ae, fe, and CLr of GSK2251052 as data permit. | within 14 days of first dose

SECONDARY OUTCOMES:
AUC(0-t), AUC(0-inf), and Cmax following single dose administration for the assessment of dose proportionality | within 72 h of dosing
Trough plasma concentrations | within 10 days of first dose
Accumulation based on AUC(Ro) and Cmax (RCmax) and determine the steady-state ratio (Rss) | within 14 days of first dose
AUC(0-t)am and Cmax,am following repeat administration at different doses for the assessment of dose proportionality | within 14 days of first dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

REFERENCES:
- See also: Results for study 114470 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114470?search=study&search_terms=114470#rs